CLINICAL TRIAL: NCT02335762
Title: Dietary Intake of Conjugated Linoleic Acid in a Cohort of Healthy Students in Italy
Brief Title: Dietary Conjugated Linoleic Acid (CLA) Intake Among Students in Italy
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Filippo Rossi, Researcher, Catholic University of the Sacred Heart
Other Study IDs: 24475/14
Record Dates: First submitted 2014-12-15; First posted 2015-01-12 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: CLA Intake From Different Food Sources

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
40 healthy subjects were recruited using advertisements posted at the Catholic University of Piacenza, between January and October 2012. Height (using a stadiometer) and weight (using a Gima scale) of each subject were measured and the body mass index (BMI) was calculated (kg/m2). Subjects who satisfied inclusion criteria were instructed on how to document all food and drink consumed daily for 3 days using a diary previously used in the Italian National Survey INRAN-SCAI. They were asked to eat as usual in subsequent 3 days to emulate as best their habits. They were educated to report also the place, time, number and quantity of serving portions consumed. If they were not able to weight exactly each portion, a photographic atlas developed for the Italian component of the European Prospective Investigation into Cancer and Nutrition (EPIC) study was used. At the end of the three days the food diaries were checked and for each subject the energy intake was estimated.

ELIGIBILITY:
Inclusion Criteria:

* self-reported healthy
* not suffering disorders of lipid metabolism and from eating disorders.

Exclusion Criteria:

* pregnant or breast-feeding,
* subjects consuming an energy-restricted diet
* vegan or vegetarians.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 40 healthy students
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
CLA intake (food questionnaire crossed with data on CLA amount in foods) | 3 days
  food questionnaire crossed with data on CLA amount in foods